CLINICAL TRIAL: NCT04206891
Title: Understanding How CDH1 Germline Mutations Affect Hereditary Lobular Breast Cancer
Brief Title: CDH1 Germline Mutations in Lobular Breast Cancer
Status: Completed | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 0834/
Record Dates: First submitted 2019-04-04; First posted 2019-12-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Lobular Breast Carcinoma; CDH1 Gene Inactivation
MeSH Terms: conditions — Carcinoma, Lobular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Bilateral lobular invasive breast cancer
- Group 2: Invasive lobular breast cancer with age at onset <= 45 years
- Group 3: Invasive lobular breast cancer with family history for breast cancer
- Group 4: In situ lobular breast cancer with age at onset <= 45 years
- Group 5: In situ lobular breast cancer with family history for breast cancer

SUMMARY:
Invasive lobular breast carcinoma (ILBC) represents 5-15% of all invasive BCs. The CDH1 gene (OMIM no. 192090), located on the chromosome 16q22.1, encodes for the E-cadherin protein, a key regulator of cell adhesion. Loss of E-cadherin expression is frequently detected in LBC CDH1 germline loss-of-function mutations are associated with the autosomal dominant cancer-predisposition syndrome, hereditary diffuse gastric cancer (HDGC; OMIM no. 137215). The cumulative risk of LBC for women with a CDH1 mutation is estimated to be 42% (95% CI 23% to 68%) by 80 years, when it is a component of HDGC syndrome.

Recently, some authors described CDH1 germline mutations in women with in situ or ILBC with early onset (<45 or <50) and bilateral in situ or ILBC with no family history of HDGC. These results are opening a new scenario, suggesting that CDH1 could be a susceptibility gene for LBC in women without a family history of DGC.

The first aim of this study is to investigate prevalence of CDH1 in this specific population of women with early onset (<45 or <50) in situ or ILBC, bilateral LBC or LBC with no family history of HDGC.

DETAILED DESCRIPTION:
Invasive lobular breast carcinoma (ILBC) represents 5-15% of all invasive BCs. LBC presents relevant differences in the transcriptomic profiles, metastatic pattern, and clinical behaviour compared to infiltrating ductal BC.

The CDH1 gene (OMIM no. 192090), located on the chromosome 16q22.1, encodes for the E-cadherin protein, a key regulator of cell adhesion. Loss of E-cadherin expression is frequently detected in LBC.

CDH1 germline loss-of-function mutations are associated with the autosomal dominant cancer-predisposition syndrome, hereditary diffuse gastric cancer (HDGC; OMIM no. 137215). The cumulative risk of LBC for women with a CDH1 mutation is estimated to be 42% (95% CI 23% to 68%) by 80 years, when it is a component of HDGC syndrome.

Recently, updated clinical guidelines for CDH1 testing criteria have been published. For LBC, CDH1 genetic screening has been suggested for families with diagnosed of both DGC and LBC (one diagnosis before the age of 50) and patients with bilateral or familial LBC before the age of 50.

Recently, some authors described CDH1 germline mutations in women with in situ or ILBC with early onset (<45 or <50) and bilateral in situ or ILBC with no family history of HDGC. These results are opening a new scenario, suggesting that CDH1 could be a susceptibility gene for LBC in women without a family history of DGC.

The investigators have revised all literature data about early-onset LBC and CDH1 germline mutations, excluding pedigrees associated with DGCs. In detail, 482 cases of LBCs were screened for CDH1 constitutional mutations. Family history for breast carcinoma was documented in 40.7 % of the considered probands and 20.3 % presented a bilateral BC manifestation. Mean age at onset was 46 years. Fourteen novels deleterious alterations (2.9 %) have been reported; 5 were missense (35.7 %), 3 mutations affected the splicing sites (21.4 %), 3 deletions (21.4 %), 2 insertions (14.3 %) and 1 stop codon (7.2 %). These mutations affect different CDH1 gene domains, spanning almost all 16 exons and introns 1-7-13 boundaries. Two missense mutations were defined as potentially pathogenic variants in vitro and in silico analysis [Corso et al. Fam Cancer 2016]. Overall, about 3% of the screened population with LBC have a mutation.

To date, no clear-cut genetic indicators for increased risk have been identified in patients with lobular breast cancer (LBC).

The first aim of this study is to investigate prevalence of CDH1 in this specific population of women with early onset (<45 or <50) in situ or ILBC, bilateral LBC or LBC with no family history of HDGC.

The investigators hypothesize that CDH1 is a susceptibility gene for LBC and that a novel and rare syndrome (called as hereditary LBC), independent from the classic HDGC setting, should be described, especially in subjects with early onset of LBC, before 45 years at diagnosis, and in bilateral LBC manifestation.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral lobular breast cancer or Lobular breast cancer with age at onset <= 45 years or Lobular breast cancer with family history for breast cancer
* Patients with blood available in IEO biobank

Exclusion Criteria:

* Patients with a previous cancer (except for colon cancer, stomach cancer and lobular breast cancer).
* Patients with germline BRCA1/2 patogenetic mutation will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 1997 to 2016 we collected data from a total of 1544 patients with invasive LBC and 230 with in situ histotype.
  For CDH1 genetic screening, an additional population will be considered prospectively between the range 2017-2018 Among them we will have to identified patients with a BRCA1/2 pathogenetic mutation.
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Relative frequency of patients with a mutation in CDH1 germline | 6 months
  Number of patients with mutation in CDH1 germline per each group identified

SECONDARY OUTCOMES:
Frequency of patients with a mutation in CDH1 germline by disease status | 6 months
  Number of patients with a mutation in CDH1 germline stratified by disease status to investigate the prevalence of this mutation status between invasive and in situ BC
Frequency of patients with a mutation in CDH1 germline by clinical strata | 6 months
  Number of patients with a mutation in CDH1 germline stratified by clinical data to investigate the prevalence of this mutation status betweenr early onset LBC (<45 years), bilateral LBC and LBC with family history for breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Corso, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy